CLINICAL TRIAL: NCT05171205
Title: Spinal Cord Stimulation for Parkinsonism: a Single-center, Single-arm Open Trial
Brief Title: Spinal Cord Stimulation for Parkinsonism
Acronym: SCS for PDS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCS_PDS
Record Dates: First submitted 2021-11-23; First posted 2021-12-28 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-01

CONDITIONS: Parkinsonism
MeSH Terms: conditions — Parkinsonian Disorders | interventions — Spinal Cord Stimulation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Spinal cord stimulation(SCS) implantation (Experimental): Phase I:
  1. Spinal cord segment is selected as the puncture location according to the patient's symptom and the condition of the patient's spinal cord. Percutaneous puncture is performed under X-ray guidance. One or two electrodes are placed in the patient's epidural cavity, and the electrode position is adjusted intraoperatively and by the patient's feedback of the current stimulation position until the current can cover the entire area.
  2. An extension lead is connected, an external temporary stimulator is attached, and the patient decides whether to proceed to full implantation in phase II after 7-10 days of phase I testing experience.
  Phase II:
  The complete SCS system is implanted under local anesthesia or epidural anesthesia after successful testing. A subcutaneous capsular bag is usually created in the lower abdomen and the implanted electrodes are connected to the pulse generator through a connecting wire in the subcutaneous tunnel.
  Interventions: Device: Spinal cord stimulation

INTERVENTIONS:
Device: Spinal cord stimulation — Spinal cord stimulation (SCS) is a very thin electrode implanted in the dorsal epidural space of the spinal cord to improve the patient's symptoms by stimulating the spinal nerves with pulsed electrical currents, which attenuate or enhance the flow of nerve impulses from the periphery to the central system, i.e., stimulating thick fibers to achieve therapeutic results. SCS system consists of three components: an electrode implanted in the epidural space of the patient's spinal cord, a stimulator implanted subcutaneously in the abdomen or buttocks that delivers electrical impulses, and an extension cord that connects the two.

SUMMARY:
Spinal Cord Stimulation (SCS) is a newly emerged neuromodulation technique in recent years. It is now a mature technique in the treatment of chronic pain and is generally accepted by patients because of its non-destructive and reversible nature, few complications, no side effects, and avoidance of unnecessary surgical procedures. Combining the results of previous studies and the group's previous research, this study first proposes an innovative treatment protocol for PDS with SCS. We intend to conduct a prospective single-center open clinical trial to evaluate the improvement of orthostatic hypotension, urinary retention, sleep disturbance, dysarthria, and dysphagia in Parkinsonism (PDS) patients before and after SCS treatment, and shed new light on the treatment for PDS.

ELIGIBILITY:
Inclusion criteria:

1. Diagnosed with parkinsonism according to MDS clinical diagnostic criteria for Parkinson's disease
2. Aged between 50 and 80 years
3. Able and willing to follow instruction of the researcher
4. No other conditions that the researchers consider inappropriate for inclusion

Exclusion criteria:

1. Severe depression (HAMD-17 above 17 as moderate to severe) or anxiety
2. Pregnancy
3. History of alcoholism
4. Non-neurological disease-related symptoms that prevent patients from participation in the study

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of blood pressure from baseline to 3 months post-operation | 3 months
  Change of on-off delta systolic blood pressure and delta diastolic blood pressure from baseline to 3 months post-operation. Delta systolic blood pressure equals the systolic blood pressure of the patient lying minus the systolic blood pressure of the patient standing up for 10 minutes.
  Delta diastolic blood pressure equals the diastolic blood pressure of the patient lying minus the diastolic blood pressure of the patient standing up for 10 minutes.
Change of blood pressure from baseline to 6 months post-operation | 6 months
  Change of on-off delta systolic blood pressure and delta diastolic blood pressure from baseline to 6 months post-operation. Delta systolic blood pressure equals the systolic blood pressure of the patient lying minus the systolic blood pressure of the patient standing up for 10 minutes.
  Delta diastolic blood pressure equals the diastolic blood pressure of the patient lying minus the diastolic blood pressure of the patient standing up for 10 minutes.
Change of blood pressure from baseline to 9 months post-operation | 9 months
  Change of on-off delta systolic blood pressure and delta diastolic blood pressure from baseline to 9 months post-operation. Delta systolic blood pressure equals the systolic blood pressure of the patient lying minus the systolic blood pressure of the patient standing up for 10 minutes.
  Delta diastolic blood pressure equals the diastolic blood pressure of the patient lying minus the diastolic blood pressure of the patient standing up for 10 minutes.
Change of blood pressure from baseline to 12 months post-operation | 12 months
  Change of on-off delta systolic blood pressure and delta diastolic blood pressure from baseline to 12 months post-operation. Delta systolic blood pressure equals the systolic blood pressure of the patient lying minus the systolic blood pressure of the patient standing up for 10 minutes.
  Delta diastolic blood pressure equals the diastolic blood pressure of the patient lying minus the diastolic blood pressure of the patient standing up for 10 minutes.
Change of blood pressure from baseline to 18 months post-operation | 18 months
  Change of on-off delta systolic blood pressure and delta diastolic blood pressure from baseline to 18 months post-operation. Delta systolic blood pressure equals the systolic blood pressure of the patient lying minus the systolic blood pressure of the patient standing up for 10 minutes. Delta diastolic blood pressure equals the diastolic blood pressure of the patient lying minus the diastolic blood pressure of the patient standing up for 10 minutes.
Change of blood pressure from baseline to 24 months post-operation | 24 months
  Change of on-off delta systolic blood pressure and delta diastolic blood pressure from baseline to 24 months post-operation. Delta systolic blood pressure equals the systolic blood pressure of the patient lying minus the systolic blood pressure of the patient standing up for 10 minutes. Delta diastolic blood pressure equals the diastolic blood pressure of the patient lying minus the diastolic blood pressure of the patient standing up for 10 minutes.

SECONDARY OUTCOMES:
Change of oxygen desaturation index from baseline to 3 months post-operation | 3 months
  Change of oxygen desaturation index measured by on-off polysomnography from baseline to 3 months post-operation
Change of oxygen desaturation index from baseline to 6 months post-operation | 6 months
  Change of oxygen desaturation index measured by on-off polysomnography from baseline to 6 months post-operation
Change of oxygen desaturation index from baseline to 9 months post-operation | 9 months
  Change of oxygen desaturation index measured by on-off polysomnography from baseline to 9 months post-operation
Change of oxygen desaturation index from baseline to 12 months post-operation | 12 months
  Change of oxygen desaturation index measured by on-off polysomnography from baseline to 12 months post-operation
Change of oxygen desaturation index from baseline to 18 months post-operation | 18 months
  Change of oxygen desaturation index measured by on-off polysomnography from baseline to 18 months post-operation
Change of oxygen desaturation index from baseline to 24 months post-operation | 24 months
  Change of oxygen desaturation index measured by on-off polysomnography from baseline to 24 months post-operation
Change of apnea hypopnea index from baseline to 3 months post-operation | 3 months
  Change of apnea hypopnea index measured by on-off polysomnography from baseline to 3 months post-operation
Change of apnea hypopnea index from baseline to 6 months post-operation | 6 months
  Change of apnea hypopnea index measured by on-off polysomnography from baseline to 6 months post-operation
Change of apnea hypopnea index from baseline to 9 months post-operation | 9 months
  Change of apnea hypopnea index measured by on-off polysomnography from baseline to 9 months post-operation
Change of apnea hypopnea index from baseline to 12 months post-operation | 12 months
  Change of apnea hypopnea index measured by on-off polysomnography from baseline to 12 months post-operation
Change of apnea hypopnea index from baseline to 18 months post-operation | 18 months
  Change of apnea hypopnea index measured by on-off polysomnography from baseline to 18 months post-operation
Change of apnea hypopnea index from baseline to 24 months post-operation | 24 months
  Change of apnea hypopnea index measured by on-off polysomnography from baseline to 24 months post-operation
Change of on-off 24-hour blood pressure monitoring from baseline to 3 months post-operation | 3 months
  Change of on-off 24-hour blood pressure monitoring from baseline to 3 months post-operation.
Change of on-off 24-hour blood pressure monitoring from baseline to 6 months post-operation | 6 months
  Change of on-off 24-hour blood pressure monitoring from baseline to 6 months post-operation.
Change of on-off 24-hour blood pressure monitoring from baseline to 9 months post-operation | 9 months
  Change of on-off 24-hour blood pressure monitoring from baseline to 9 months post-operation.
Change of on-off 24-hour blood pressure monitoring from baseline to 12 months post-operation | 12 months
  Change of on-off 24-hour blood pressure monitoring from baseline to 12 months post-operation.
Change of on-off 24-hour blood pressure monitoring from baseline to 18 months post-operation | 18 months
  Change of on-off 24-hour blood pressure monitoring from baseline to 18 months post-operation.
Change of on-off 24-hour blood pressure monitoring from baseline to 24 months post-operation | 24 months
  Change of on-off 24-hour blood pressure monitoring from baseline to 24 months post-operation.
Change of on-off time patient spend in supine status, seated status, standing/walking status from baseline to 3 months post-operation | 3 months
  Change of on-off time patient spend in supine status, seated status, standing/walking status from baseline to 3 months post-operation.
Change of on-off time patient spend in supine status, seated status, standing/walking status from baseline to 6 months post-operation | 6 months
  Change of on-off time patient spend in supine status, seated status, standing/walking status from baseline to 6 months post-operation.
Change of on-off time patient spend in supine status, seated status, standing/walking status from baseline to 9 months post-operation | 9 months
  Change of on-off time patient spend in supine status, seated status, standing/walking status from baseline to 9 months post-operation.
Change of on-off time patient spend in supine status, seated status, standing/walking status from baseline to 12 months post-operation | 12 months
  Change of on-off time patient spend in supine status, seated status, standing/walking status from baseline to 12 months post-operation.
Change of on-off time patient spend in supine status, seated status, standing/walking status from baseline to 18 months post-operation | 18 months
  Change of on-off time patient spend in supine status, seated status, standing/walking status from baseline to 18 months post-operation.
Change of on-off time patient spend in supine status, seated status, standing/walking status from baseline to 24 months post-operation | 24 months
  Change of on-off time patient spend in supine status, seated status, standing/walking status from baseline to 24 months post-operation.
Change of serum catecholamine neurotransmitter levels from baseline to 3 months post-operation | 3 months
  Change of on-off delta serum catecholamine neurotransmitter levels from baseline to 3 months post-operation. Delta serum catecholamine neurotransmitter levels equals the serum catecholamine neurotransmitter levels of the patient lying minus the serum catecholamine neurotransmitter levels of the patient standing up for 10 minutes.
Change of serum catecholamine neurotransmitter levels from baseline to 6 months post-operation | 6 months
  Change of on-off delta serum catecholamine neurotransmitter levels from baseline to 6 months post-operation. Delta serum catecholamine neurotransmitter levels equals the serum catecholamine neurotransmitter levels of the patient lying minus the serum catecholamine neurotransmitter levels of the patient standing up for 10 minutes.
Change of serum catecholamine neurotransmitter levels from baseline to 9 months post-operation | 9 months
  Change of on-off delta serum catecholamine neurotransmitter levels from baseline to 9 months post-operation. Delta serum catecholamine neurotransmitter levels equals the serum catecholamine neurotransmitter levels of the patient lying minus the serum catecholamine neurotransmitter levels of the patient standing up for 10 minutes.
Change of serum catecholamine neurotransmitter levels from baseline to 12 months post-operation | 12 months
  Change of on-off delta serum catecholamine neurotransmitter levels from baseline to 12 months post-operation. Delta serum catecholamine neurotransmitter levels equals the serum catecholamine neurotransmitter levels of the patient lying minus the serum catecholamine neurotransmitter levels of the patient standing up for 10 minutes.
Change of serum catecholamine neurotransmitter levels from baseline to 18 months post-operation | 18 months
  Change of on-off delta serum catecholamine neurotransmitter levels from baseline to 18 months post-operation. Delta serum catecholamine neurotransmitter levels equals the serum catecholamine neurotransmitter levels of the patient lying minus the serum catecholamine neurotransmitter levels of the patient standing up for 10 minutes.
Change of serum catecholamine neurotransmitter levels from baseline to 24 months post-operation | 24 months
  Change of on-off delta serum catecholamine neurotransmitter levels from baseline to 24 months post-operation. Delta serum catecholamine neurotransmitter levels equals the serum catecholamine neurotransmitter levels of the patient lying minus the serum catecholamine neurotransmitter levels of the patient standing up for 10 minutes.
Change of on-off delta heart rate variability from baseline to 3 months post-operation | 3 months
  Change of on-off delta heart rate variability from baseline to 3 months post-operation. Delta heart rate variability equals the heart rate variability of the patient lying minus the heart rate variability of the patient standing up for 10 minutes.
Change of on-off delta heart rate variability from baseline to 6 months post-operation | 6 months
  Change of on-off delta heart rate variability from baseline to 6 months post-operation. Delta heart rate variability equals the heart rate variability of the patient lying minus the heart rate variability of the patient standing up for 10 minutes.
Change of on-off delta heart rate variability from baseline to 9 months post-operation | 9 months
  Change of on-off delta heart rate variability from baseline to 9 months post-operation. Delta heart rate variability equals the heart rate variability of the patient lying minus the heart rate variability of the patient standing up for 10 minutes.
Change of on-off delta heart rate variability from baseline to 12 months post-operation | 12 months
  Change of on-off delta heart rate variability from baseline to 12 months post-operation. Delta heart rate variability equals the heart rate variability of the patient lying minus the heart rate variability of the patient standing up for 10 minutes.
Change of on-off delta heart rate variability from baseline to 18 months post-operation | 18 months
  Change of on-off delta heart rate variability from baseline to 18 months post-operation. Delta heart rate variability equals the heart rate variability of the patient lying minus the heart rate variability of the patient standing up for 10 minutes.
Change of on-off delta heart rate variability from baseline to 24 months post-operation | 24 months
  Change of on-off delta heart rate variability from baseline to 24 months post-operation. Delta heart rate variability equals the heart rate variability of the patient lying minus the heart rate variability of the patient standing up for 10 minutes.
Change of length of walking during 6-minute walking test from baseline to 3 months post-operation | 3 months
  Change of on-off length of walking during 6-minute walking test from baseline to 3 months post-operation.
Change of length of walking during 6-minute walking test from baseline to 6 months post-operation | 6 months
  Change of on-off length of walking during 6-minute walking test from baseline to 6 months post-operation.
Change of length of walking during 6-minute walking test from baseline to 9 months post-operation | 9 months
  Change of on-off length of walking during 6-minute walking test from baseline to 9 months post-operation.
Change of length of walking during 6-minute walking test from baseline to 12 months post-operation | 12 months
  Change of on-off length of walking during 6-minute walking test from baseline to 12 months post-operation.
Change of length of walking during 6-minute walking test from baseline to 18 months post-operation | 18 months
  Change of on-off length of walking during 6-minute walking test from baseline to 18 months post-operation.
Change of length of walking during 6-minute walking test from baseline to 24 months post-operation | 24 months
  Change of on-off length of walking during 6-minute walking test from baseline to 24 months post-operation.
Change of time of walking during 6-minute walking test from baseline to 3 months post-operation | 3 months
  Change of on-off time of walking during 6-minute walking test from baseline to 3 months post-operation.
Change of time of walking during 6-minute walking test from baseline to 6 months post-operation | 6 months
  Change of on-off time of walking during 6-minute walking test from baseline to 6 months post-operation.
Change of time of walking during 6-minute walking test from baseline to 9 months post-operation | 9 months
  Change of on-off time of walking during 6-minute walking test from baseline to 9 months post-operation.
Change of time of walking during 6-minute walking test from baseline to 12 months post-operation | 12 months
  Change of on-off time of walking during 6-minute walking test from baseline to 12 months post-operation.
Change of time of walking during 6-minute walking test from baseline to 18 months post-operation | 18 months
  Change of on-off time of walking during 6-minute walking test from baseline to 18 months post-operation.
Change of time of walking during 6-minute walking test from baseline to 24 months post-operation | 24 months
  Change of on-off time of walking during 6-minute walking test from baseline to 24 months post-operation.
Change of on-off numbers of mistakes made during Stroop Color and Word Test from baseline to 3 months post-operation | 3 months
  Change of on-off numbers of mistakes made during Stroop Color and Word Test from baseline to 3 months post-operation.
Change of on-off numbers of mistakes made during Stroop Color and Word Test from baseline to 6 months post-operation | 6 months
  Change of on-off numbers of mistakes made during Stroop Color and Word Test from baseline to 6 months post-operation.
Change of on-off numbers of mistakes made during Stroop Color and Word Test from baseline to 9 months post-operation | 9 months
  Change of on-off numbers of mistakes made during Stroop Color and Word Test from baseline to 9 months post-operation.
Change of on-off numbers of mistakes made during Stroop Color and Word Test from baseline to 12 months post-operation | 12 months
  Change of on-off numbers of mistakes made during Stroop Color and Word Test from baseline to 12 months post-operation.
Change of on-off numbers of mistakes made during Stroop Color and Word Test from baseline to 18 months post-operation | 18 months
  Change of on-off numbers of mistakes made during Stroop Color and Word Test from baseline to 18 months post-operation.
Change of on-off numbers of mistakes made during Stroop Color and Word Test from baseline to 24 months post-operation | 24 months
  Change of on-off numbers of mistakes made during Stroop Color and Word Test from baseline to 24 months post-operation.
Change of on-off time to complete the Stroop Color and Word Test from baseline to 3 months post-operation | 3 months
  Change of on-off time to complete the Stroop Color and Word Test from baseline to 3 months post-operation.
Change of on-off time to complete the Stroop Color and Word Test from baseline to 6 months post-operation | 6 months
  Change of on-off time to complete the Stroop Color and Word Test from baseline to 6 months post-operation.
Change of on-off time to complete the Stroop Color and Word Test from baseline to 9 months post-operation | 9 months
  Change of on-off time to complete the Stroop Color and Word Test from baseline to 9 months post-operation.
Change of on-off time to complete the Stroop Color and Word Test from baseline to 12 months post-operation | 12 months
  Change of on-off time to complete the Stroop Color and Word Test from baseline to 12 months post-operation.
Change of on-off time to complete the Stroop Color and Word Test from baseline to 18 months post-operation | 18 months
  Change of on-off time to complete the Stroop Color and Word Test from baseline to 18 months post-operation.
Change of on-off time to complete the Stroop Color and Word Test from baseline to 24 months post-operation | 24 months
  Change of on-off time to complete the Stroop Color and Word Test from baseline to 24 months post-operation.
Change of on-off delta brain cortex oxygenated hemoglobin levels from baseline to 3 months post-operation | 3 months
  Change of on-off delta brain cortex oxygenated hemoglobin levels from baseline to 3 months post-operation. Delta brain cortex oxygenated hemoglobin levels equals the brain cortex oxygenated hemoglobin levels of the patient lying minus the brain cortex oxygenated hemoglobin levels of the patient standing up for 10 minutes.
Change of on-off delta brain cortex oxygenated hemoglobin levels from baseline to 6 months post-operation | 6 months
  Change of on-off delta brain cortex oxygenated hemoglobin levels from baseline to 6 months post-operation. Delta brain cortex oxygenated hemoglobin levels equals the brain cortex oxygenated hemoglobin levels of the patient lying minus the brain cortex oxygenated hemoglobin levels of the patient standing up for 10 minutes.
Change of on-off delta brain cortex oxygenated hemoglobin levels from baseline to 9 months post-operation | 9 months
  Change of on-off delta brain cortex oxygenated hemoglobin levels from baseline to 9 months post-operation. Delta brain cortex oxygenated hemoglobin levels equals the brain cortex oxygenated hemoglobin levels of the patient lying minus the brain cortex oxygenated hemoglobin levels of the patient standing up for 10 minutes.
Change of on-off delta brain cortex oxygenated hemoglobin levels from baseline to 12 months post-operation | 12 months
  Change of on-off delta brain cortex oxygenated hemoglobin levels from baseline to 12 months post-operation. Delta brain cortex oxygenated hemoglobin levels equals the brain cortex oxygenated hemoglobin levels of the patient lying minus the brain cortex oxygenated hemoglobin levels of the patient standing up for 10 minutes.
Change of on-off delta brain cortex oxygenated hemoglobin levels from baseline to 18 months post-operation | 18 months
  Change of on-off delta brain cortex oxygenated hemoglobin levels from baseline to 18 months post-operation. Delta brain cortex oxygenated hemoglobin levels equals the brain cortex oxygenated hemoglobin levels of the patient lying minus the brain cortex oxygenated hemoglobin levels of the patient standing up for 10 minutes.
Change of on-off delta brain cortex oxygenated hemoglobin levels from baseline to 24 months post-operation | 24 months
  Change of on-off delta brain cortex oxygenated hemoglobin levels from baseline to 24 months post-operation. Delta brain cortex oxygenated hemoglobin levels equals the brain cortex oxygenated hemoglobin levels of the patient lying minus the brain cortex oxygenated hemoglobin levels of the patient standing up for 10 minutes.
Change of dysarthria symptom from baseline to 3 months post-operation | 3 months
  Change of dysarthria symptom measured by on-off Dysphonia Severity Index of Atoms Speech Assessment System from baseline to 3 months post-operation
Change of dysarthria symptom from baseline to 6 months post-operation | 6 months
  Change of dysarthria symptom measured by on-off Dysphonia Severity Index of Atoms Speech Assessment System from baseline to 6 months post-operation
Change of dysarthria symptom from baseline to 9 months post-operation | 9 months
  Change of dysarthria symptom measured by on-off Dysphonia Severity Index of Atoms Speech Assessment System from baseline to 9 months post-operation
Change of dysarthria symptom from baseline to 12 months post-operation | 12 months
  Change of dysarthria symptom measured by on-off Dysphonia Severity Index of Atoms Speech Assessment System from baseline to 12 months post-operation
Change of dysarthria symptom from baseline to 18 months post-operation | 18 months
  Change of dysarthria symptom measured by on-off Dysphonia Severity Index of Atoms Speech Assessment System from baseline to 18 months post-operation
Change of dysarthria symptom from baseline to 24 months post-operation | 24 months
  Change of dysarthria symptom measured by on-off Dysphonia Severity Index of Atoms Speech Assessment System from baseline to 24 months post-operation
Change of urinary retention from baseline to 3 months post-operation | 3 months
  The change of volume of urinary retention measured by ultrasound and urodynamic study from baseline to 3 months post-operation
Change of urinary retention from baseline to 6 months post-operation | 6 months
  The change of volume of urinary retention measured by ultrasound and urodynamic study from baseline to 6 months post-operation
Change of urinary retention from baseline to 9 months post-operation | 9 months
  The change of volume of urinary retention measured by ultrasound and urodynamic study from baseline to 9 months post-operation
Change of urinary retention from baseline to 12 months post-operation | 12 months
  The change of volume of urinary retention measured by ultrasound and urodynamic study from baseline to 12 months post-operation
Change of urinary retention from baseline to 18 months post-operation | 18 months
  The change of volume of urinary retention measured by ultrasound and urodynamic study from baseline to 18 months post-operation
Change of urinary retention from baseline to 24 months post-operation | 24 months
  The change of volume of urinary retention measured by ultrasound and urodynamic study from baseline to 24 months post-operation
Change of MDS-UPDRS from baseline to 3 months post-operation | 3 months
  The change of on- off rating of the Movement Disorders Society sponsored Unified Parkinson's Disease Rating Scale (MDS-UPDRS) from baseline to 3 months post-operation
Change of MDS-UPDRS from baseline to 6 months post-operation | 6 months
  The change of on- off rating of the Movement Disorders Society sponsored Unified Parkinson's Disease Rating Scale (MDS-UPDRS) from baseline to 6 months post-operation
Change of MDS-UPDRS from baseline to 9 months post-operation | 9 months
  The change of on- off rating of the Movement Disorders Society sponsored Unified Parkinson's Disease Rating Scale (MDS-UPDRS) from baseline to 9 months post-operation
Change of MDS-UPDRS from baseline to 12 months post-operation | 12 months
  The change of on- off rating of the Movement Disorders Society sponsored Unified Parkinson's Disease Rating Scale (MDS-UPDRS) from baseline to 12 months post-operation
Change of MDS-UPDRS from baseline to 18 months post-operation | 18 months
  The change of on- off rating of the Movement Disorders Society sponsored Unified Parkinson's Disease Rating Scale (MDS-UPDRS) from baseline to 18 months post-operation
Change of MDS-UPDRS from baseline to 24 months post-operation | 24 months
  The change of on- off rating of the Movement Disorders Society sponsored Unified Parkinson's Disease Rating Scale (MDS-UPDRS) from baseline to 24 months post-operation
Change of UMSARS from baseline to 3 months post-operation | 3 months
  The change of on- off rating of the Unified Multiple System Atrophy Rating Scale (UMSARS) from baseline to 3 months post-operation
Change of UMSARS from baseline to 6 months post-operation | 6 months
  The change of on- off rating of the Unified Multiple System Atrophy Rating Scale (UMSARS) from baseline to 6 months post-operation
Change of UMSARS from baseline to 9 months post-operation | 9 months
  The change of on- off rating of the Unified Multiple System Atrophy Rating Scale (UMSARS) from baseline to 9 months post-operation
Change of UMSARS from baseline to 12 months post-operation | 12 months
  The change of on- off rating of the Unified Multiple System Atrophy Rating Scale (UMSARS) from baseline to 12 months post-operation
Change of UMSARS from baseline to 18 months post-operation | 18 months
  The change of on- off rating of the Unified Multiple System Atrophy Rating Scale (UMSARS) from baseline to 18 months post-operation
Change of UMSARS from baseline to 24 months post-operation | 24 months
  The change of on- off rating of the Unified Multiple System Atrophy Rating Scale (UMSARS) from baseline to 24 months post-operation
Change of lowest oxygen saturation from baseline to 3 months post-operation | 3 months
  Change of lowest oxygen saturation measured by on-off polysomnography from baseline to 3 months post-operation
Change of lowest oxygen saturation from baseline to 6 months post-operation | 6 months
  Change of lowest oxygen saturation measured by on-off polysomnography from baseline to 6 months post-operation
Change of lowest oxygen saturation from baseline to 9 months post-operation | 9 months
  Change of lowest oxygen saturation measured by on-off polysomnography from baseline to 9 months post-operation
Change of lowest oxygen saturation from baseline to 12 months post-operation | 12 months
  Change of lowest oxygen saturation measured by on-off polysomnography from baseline to 12 months post-operation
Change of lowest oxygen saturation from baseline to 18 months post-operation | 18 months
  Change of lowest oxygen saturation measured by on-off polysomnography from baseline to 18 months post-operation
Change of lowest oxygen saturation from baseline to 24 months post-operation | 24 months
  Change of lowest oxygen saturation measured by on-off polysomnography from baseline to 24 months post-operation
Change of mean oxygen saturation from baseline to 3 months post-operation | 3 months
  Change of mean oxygen saturation measured by on-off polysomnography from baseline to 3 months post-operation
Change of mean oxygen saturation from baseline to 6 months post-operation | 6 months
  Change of mean oxygen saturation measured by on-off polysomnography from baseline to 6 months post-operation
Change of mean oxygen saturation from baseline to 9 months post-operation | 9 months
  Change of mean oxygen saturation measured by on-off polysomnography from baseline to 9 months post-operation
Change of mean oxygen saturation from baseline to 12 months post-operation | 12 months
  Change of mean oxygen saturation measured by on-off polysomnography from baseline to 12 months post-operation
Change of mean oxygen saturation from baseline to 18 months post-operation | 18 months
  Change of mean oxygen saturation measured by on-off polysomnography from baseline to 18 months post-operation
Change of mean oxygen saturation from baseline to 24 months post-operation | 24 months
  Change of mean oxygen saturation measured by on-off polysomnography from baseline to 24 months post-operation
Change of SCOPA-AUT from baseline to 3 months post-operation | 3 months
  Change of scales for outcomes in Parkinson's disease - autonomic dysfunction from baseline to 3 months post-operation
Change of SCOPA-AUT from baseline to 6 months post-operation | 6 months
  Change of scales for outcomes in Parkinson's disease - autonomic dysfunction from baseline to 6 months post-operation
Change of SCOPA-AUT from baseline to 9 months post-operation | 9 months
  Change of scales for outcomes in Parkinson's disease - autonomic dysfunction from baseline to 9 months post-operation
Change of SCOPA-AUT from baseline to 12 months post-operation | 12 months
  Change of scales for outcomes in Parkinson's disease - autonomic dysfunction from baseline to 12 months post-operation
Change of SCOPA-AUT from baseline to 18 months post-operation | 18 months
  Change of scales for outcomes in Parkinson's disease - autonomic dysfunction from baseline to 18 months post-operation
Change of SCOPA-AUT from baseline to 24 months post-operation | 24 months
  Change of scales for outcomes in Parkinson's disease - autonomic dysfunction from baseline to 24 months post-operation
Change of delta cerebral artery velocity from baseline to 3 months post-operation | 3 months
  Change of on-off delta cerebral artery velocity from baseline to 3 months post-operation. Delta cerebral artery velocity equals cerebral artery velocity of the patient lying minus the systolic blood pressure of the patient standing up for 10 minutes.
Change of delta cerebral artery velocity from baseline to 6 months post-operation | 6 months
  Change of on-off delta cerebral artery velocity from baseline to 6 months post-operation. Delta cerebral artery velocity equals cerebral artery velocity of the patient lying minus the systolic blood pressure of the patient standing up for 10 minutes.
Change of delta cerebral artery velocity from baseline to 9 months post-operation | 9 months
  Change of on-off delta cerebral artery velocity from baseline to 9 months post-operation. Delta cerebral artery velocity equals cerebral artery velocity of the patient lying minus the systolic blood pressure of the patient standing up for 10 minutes.
Change of delta cerebral artery velocity from baseline to 12 months post-operation | 12 months
  Change of on-off delta cerebral artery velocity from baseline to 12 months post-operation. Delta cerebral artery velocity equals cerebral artery velocity of the patient lying minus the systolic blood pressure of the patient standing up for 10 minutes.
Change of delta cerebral artery velocity from baseline to 18 months post-operation | 18 months
  Change of on-off delta cerebral artery velocity from baseline to 18 months post-operation. Delta cerebral artery velocity equals cerebral artery velocity of the patient lying minus the systolic blood pressure of the patient standing up for 10 minutes.
Change of delta cerebral artery velocity from baseline to 24 months post-operation | 24 months
  Change of on-off delta cerebral artery velocity from baseline to 24 months post-operation. Delta cerebral artery velocity equals cerebral artery velocity of the patient lying minus the systolic blood pressure of the patient standing up for 10 minutes.
Change of TUG from baseline to 3 months post-operation | 3 months
  Change of on-off timed up and go from baseline to 3 months post-operation.
Change of TUG from baseline to 6 months post-operation | 6 months
  Change of on-off timed up and go from baseline to 6 months post-operation.
Change of TUG from baseline to 9 months post-operation | 9 months
  Change of on-off timed up and go from baseline to 9 months post-operation.
Change of TUG from baseline to 12 months post-operation | 12 months
  Change of on-off timed up and go from baseline to 12 months post-operation.
Change of TUG from baseline to 18 months post-operation | 18 months
  Change of on-off timed up and go from baseline to 18 months post-operation.
Change of TUG from baseline to 24 months post-operation | 24 months
  Change of on-off timed up and go from baseline to 24 months post-operation.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Liu, MD,PhD, Principal Investigator — Ruijin Hospital
Locations (1):
- Department of Neurology and Institute of Neurology, Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No